CLINICAL TRIAL: NCT06611917
Title: Comparative Diagnostic Values of Physical Examination Tests and Ultrasonographic Measurements in Predicting Difficult Airways
Brief Title: Diagnostic Values of Physical Examination and Ultrasonographic Measurements in Predicting Difficult Airways
Status: Completed | Type: Observational
Sponsor: Çanakkale Onsekiz Mart University (Other)
Responsible Party: Principal Investigator, Ayse Ezgi SUBASI, Specialist Doctor, Çanakkale Onsekiz Mart University
Other Study IDs: COMU-SBF-AES-01
Record Dates: First submitted 2024-07-12; First posted 2024-09-25 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-07

CONDITIONS: Airway Complication of Anesthesia
Keywords: Airway Management; Endotracheal Intubation; Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Ultrasonographic and Physical Examination Cohort: Participants in this study are patients scheduled for surgery under general anesthesia. The participants will undergo standard physical examination tests conducted by anesthesiologists before surgery and will also receive ultrasonographic measurements of the subglottic and other critical airway structures. The participants will be categorized as an observational cohort in which the ultrasonographic assessments will be compared with the results of the physical examination. The primary objective of this study is to compare the effectiveness of these two methods in predicting difficult airways.

SUMMARY:
This study evaluates the effectiveness of ultrasonographic measurements compared to traditional physical examination tests in predicting difficult airways. With no definitive gold standard for anticipating airway challenges, this research explores the diagnostic capabilities of newer, non-invasive techniques like ultrasonography-which is gaining popularity due to its ease of use and widespread availability-in the field of anesthesia. The study focuses on defining highly sensitive and easy-to-use ultrasonographic markers that could aid anesthesiologists, intensive care specialists, and emergency physicians in effective airway management.

DETAILED DESCRIPTION:
Anesthesiologists, intensive care specialists, and emergency physicians frequently encounter the challenge of managing difficult airways, a critical competency as failure to secure the airway can lead to severe consequences, including brain damage or death. Intubation, a complex procedure involving several anatomical maneuvers, has traditionally relied on physical examination indicators such as dental and facial anatomy, Mallampati score, and neck mobility to predict potential difficulties. However, these methods, while useful, often lack the accuracy needed for reliable prediction, leading to a significant percentage of unexpected difficult intubations.

Recent advances in medical imaging propose the use of radiological and ultrasonographic assessments to enhance predictive accuracy. Ultrasonography, in particular, offers a non-invasive, easily accessible method for examining airway structures, which could potentially transform standard practices in airway management. The American Society of Anesthesiologists recognizes the promising role of ultrasound in airway assessment, yet acknowledges the need for more standardized approaches to its implementation.

This research aims to compare the predictive value of physical examination findings with that of ultrasonographic measurements such as the distance from skin to hyoid bone, skin to epiglottis, and tongue volume. By establishing more reliable and sensitive ultrasonographic markers, this study seeks to provide clinicians with better tools for assessing the risk of difficult airways, ultimately contributing to safer anesthesia practices and reducing the incidence of intubation-related complications.

ELIGIBILITY:
Inclusion Criteria:

* Patients classified as American Society of Anesthesiologists (ASA) class I-II-III.
* Individuals aged between 18 and 60 years.
* Patients scheduled for elective surgery require endotracheal intubation under general anesthesia

Exclusion Criteria:

* Patients with pathologies in the airway or head and neck area (masses, cancer, congenital anomalies, acquired anatomical disorders).
* Individuals with active infections.
* Those with cervical vertebral damage.
* Patients with a history of head and neck trauma.
* Individuals who have undergone previous head and neck surgery.
* Patients with a history of head and neck radiotherapy.
* Pregnant individuals.
* Obese patients (body mass index > 30).
* Non-cooperative patients.
* Patients are requiring surgery under emergency conditions.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients aged 18-60 years undergoing surgery under general anesthesia with an ASA classification of 1-3.
Sampling Method: Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Effectiveness of Difficult Airway Prediction | up to one hour
  The primary outcome measures the effectiveness of ultrasonography and physical examination in predicting difficult airways in patients undergoing general anesthesia. Occurrence of a difficult airway is the primary outcome. A difficult airway is defined by specific clinical criteria:
  More than two intubation attempts, Intubation time exceeding 10 minutes, or Cormack-Lehane laryngoscopy grade of 3 or 4. Data will be collected during the intubation process. Intubation attempts and time will be recorded by the anesthesiologist, while the Cormack-Lehane grading will be assessed based on the view of the glottis during laryngoscopy.
  Measurement Process:
  Ultrasonographic measurements of the airway will be taken preoperatively using non-invasive ultrasound techniques. Additionally, physical examination tests will be performed preoperatively to assess airway risk. The outcome is categorized as difficult airway (yes/no) based on whether the patient meets any of the defined criteria.

CONTACTS AND LOCATIONS:
Locations (1):
- Canakkale Onsekiz Mart University, Çanakkale, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No